CLINICAL TRIAL: NCT03494647
Title: Comparison of Braces for Treatment of Sever's Disease in Barefoot Athletes
Brief Title: Comparison of Braces for Treatment of Sever's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-0611
Record Dates: First submitted 2018-03-22; First posted 2018-04-11 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Sever's Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cheetah Heel Cup (Active Comparator): Subjects randomly assigned to this group will receive the Cheetah Heel Cup at their initial visit.
  Interventions: Device: Cheetah Heel Cup
- The X Brace (Active Comparator): Subjects randomly assigned to this group will receive the X Brace at their initial visit.
  Interventions: Device: The X Brace

INTERVENTIONS:
Device: Cheetah Heel Cup — The Cheetah Heel Cup is composed of a rubber waffle that cups the athlete's heel, secured in place by a neoprene sleeve.
  Arms: Cheetah Heel Cup
Device: The X Brace — The X Brace is composed of one thick elastic band that is wrapped around the athlete's arch of the foot. A second band is wrapped around the back of the heel, crossed under the foot, and secured to the thicker band on the bottom of the foot.
  Arms: The X Brace

SUMMARY:
This study is to learn more about braces that may help young athletes diagnosed with Sever's disease. Young athletes with this diagnosis who are seen by a Sports Medicine doctor will be asked it they want to be a part of the study. Patients who want to be in the study will be randomly assigned to wear one of two kinds of braces to treat their foot pain via randomization scheme independently created by a statistician. The subjects will be given the brace for free. The subjects will also answer survey questions about the brace when they first see the doctor, then at one, two, and three months after their first visit. Data collected in this study will help doctors gain a better understanding of how to treat young athletes who do sports without shoes who are diagnosed with Sever's disease.

DETAILED DESCRIPTION:
It is widely accepted and scientifically confirmed that physical activity improves child health with positive effects on adiposity, musculoskeletal health and fitness, and cardiovascular health. Beyond the health benefits of physical activity alone, participation in sports at this crucial age enhances psychological and social health outcomes. Athletes with Sever's symptoms are limited in their ability to participate in physical activity and athletics, and it is suggested that active intervention in the management of Sever's is most appropriate to improve quality of life and outcomes without substantial time lost from sport or physical activity. Therefore, efficient and effective treatment is essential, especially for active and competitive athletes.

Standard treatment for Sever's disease is placement of heel cups in shoes and stretching or physical therapy. These interventions are effective in reducing Sever's patients' heel pain. A retrospective study showed that with treatment with a heel cup or other foot orthoses, symptoms improved within 2 months. However, there remains a distinct lack of randomized control trials evaluating treatments for Sever's in the literature. For the many young athletes with Sever's who participate in barefoot sports such as gymnastics, dance, or tae kwan do, the standard treatment is inadequate. They cannot use the recommended heel cups, which are placed in an athletic shoe. Currently, two braces are commonly used for barefoot athletes with Sever's: Cheetah Heel Cups and The X Brace. Neither of these braces are currently FDA approved as they are not considered medical devices and are marketed as an insert. Health care providers often recommend barefoot athletes purchase these braces, but no published studies evaluating their effectiveness exist in the established literature. This study will compare these two braces in an investigator-blinded, randomized control trial in order to contribute to the understanding of standard treatment for barefoot athletes with Sever's disease and improve patient outcomes by affecting clinical practice. In light of the paucity of information on and the importance of optimizing patient outcomes to improve quality of life and maintain an active lifestyle for young barefoot athletes, this prospective, randomized treatment study will compare the effectiveness of two braces in decreasing pain severity in barefoot athletes diagnosed with Sever's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-14 years
2. Participate in barefoot sports including: martial arts, dance, gymnastics, or acrobatics
3. Clinical diagnosis of Sever's or calcaneal apophysitis

Exclusion Criteria:

1. History of foot/ankle surgery
2. History of rheumatologic diagnoses
3. Prisoners,
4. pregnant females,
5. Individuals with limited decision-making capacity

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Stuart, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No sharing. Data is stored in RedCAP and will only be available for listed authors.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cheetah Heel Cup | The X Brace
Started | 21 | 22
Completed | 16 | 16
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data was only collected for participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cheetah Heel Cup | The X Brace | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (1.6) | 10.1 (1.6) | 10.4 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 11 | 11 | 22
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Height [Mean (Standard Deviation); unit: cm] | 138.2 (10.7) | 138.6 (9.0) | 138.4 (10)
Weight [Mean (Standard Deviation); unit: kg] | 32.7 (7.6) | 31.4 (5.2) | 32.05 (6.4)
Diagnosed with Seber's disease [Count of Participants; unit: Participants] | 3 | 5 | 8
Days from consent signed to beginning use of brace [Mean (Standard Deviation); unit: Days] | 6.8 (4.2) | 5.1 (3.9) | 5.95 (4.05)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) Scores
Description: The OxAFQ-C is used to measure subjective well-being for child patients (aged 5-16) affected by foot and ankle conditions using issues that are considered important to children. There are three domains to the OxAFQ-C: physical, school and play, and emotional well-being. The investigators will calculate the difference in OxAFQ-C Scores which range from 0 to 100 with higher scores indicating better functioning and higher well-being.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cheetah Heel Cup | The X Brace
Number analyzed (Participants) | 16 | 16
score on a scale
  Physical | 0.27 (0.22) | 0.22 (0.18)
  School and play | 0.19 (0.19) | 0.18 (0.25)
  Emotional wellbeing | 0.13 (0.08) | 0.05 (0.11)

2. Secondary Outcome: Changes in the Visual Analog Scale Pain Score
Description: The Visual Analog Scale pain score is on a scale from 0 (no pain) to 100 (most severe pain). The investigators will calculate the difference in Visual Analog Scale Pain Scores.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cheetah Heel Cup | The X Brace
Number analyzed (Participants) | 16 | 16
score on a scale
  At rest | -9.5 (23.1) | -7.4 (14.5)
  Daily living activities | -25.4 (30.3) | -23.6 (23.2)
  During sports | -42.4 (30.5) | -36.1 (25.8)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Cheetah Heel Cup | The X Brace
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 1/21 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cheetah Heel Cup (N=21) | The X Brace (N=22)
Heel pain with brace (Product Issues) | 1 (1) | 0 (0) — Waffle pattern in heel cup of brace was uncomfortable to participant during beginning of use.
No improvement in pain with brace (Product Issues) | 0 (0) | 1 (1) — Patient reported no improvement with brace and discontinued from the study to try another brace.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03494647/Prot_SAP_000.pdf